CLINICAL TRIAL: NCT03454997
Title: Adapting an Evidenced-based Weight Management Intervention and Testing Strategies to Increase Implementation in Community Mental Health Programs
Acronym: ACHIEVE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00156866
Record Dates: First submitted 2018-02-13; First posted 2018-03-06 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Implementation Intervention (Active Comparator): The standard version will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice as well as organizational strategy meetings.
  Interventions: Other: training including in-person and online; Other: organizational strategy meetings
- Enhanced Implementation Intervention (Active Comparator): The enhanced version will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice as well as organizational strategy meetings. The enhanced version will also include performance coaching.
  Interventions: Other: training including in-person and online; Other: organizational strategy meetings; Other: performance coaching

INTERVENTIONS:
Other: training including in-person and online — training, motivational interviewing practice
Other: organizational strategy meetings — meetings with leadership to optimize implementation of evidence-based practices
Other: performance coaching — to enhance ability to deliver the weight management intervention
  Arms: Enhanced Implementation Intervention

SUMMARY:
This is a pilot randomized clinical trial testing an implementation intervention to support delivery of a behavioral weight loss program at community mental health programs.

DETAILED DESCRIPTION:
This is a pilot randomized clinical trial testing an implementation intervention to support delivery of a behavioral weight loss program at community mental health programs. Investigators will conduct a pilot trial testing a standard and an enhanced implementation intervention. The evidenced based intervention investigators are basing the behavioral weight loss program on is ACHIEVE, and investigators are calling the translated weight loss program ACHIEVE-D. The standard version of the implementation intervention, which will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice, as well as organizational strategy meetings. The enhanced implementation intervention will include all of these strategies + performance coaching for ACHIEVE-D coaches.

ELIGIBILITY:
Coaches -

* Adult staff or peer at community mental health program
* Willing and able to participate in training and delivery of intervention

Consumers-

Inclusion Criteria:

* Age 18 and older
* Enrolled in a psychiatric rehabilitation program
* BMI ≥ 25 kg/m2
* Willing to make changes in diet and exercise to lose weight
* Willing to attend the ACHIEVE group sessions virtually or in-person at least once per week
* Ability to use a computer or tablet
* Competent and willing to give informed oral consent
* Completion of baseline data collection

Exclusion Criteria:

* Any underlying medical conditions that could seriously reduce life expectancy, ability to participate in the study, or for which dietary change/physical activity/weight loss may be contraindicated e.g., Lung disease requiring supplemental oxygen Liver failure History of anorexia nervosa or bulimia Stage V kidney disease on dialysis Cardiovascular event in the last 6 months including unstable angina, myocardial infarction, congestive heart failure, transient ischemic attack, or stroke
* Insulin dependent diabetes
* Inability to walk unassisted (e.g., uses a cane, walker, etc)
* Pregnant, breastfeeding, or planning a pregnancy during study period
* Prior or planned bariatric surgery
* Use of a prescription anti-obesity medication or over-the-counter orlistat within the past 3 months
* Self-reported weight loss of >20 lbs in the last 3 months
* Active substance use disorder, alcohol use disorder, or problem drinking (more than 14 drinks per week for women, more than 21 drinks per week for men)
* Planning to leave mental health program or move out of geographic area within 12 months
* Weight greater than 440 pounds (so as not to exceed capacity of study scale)
* Investigator judgment (e.g., for concerns over safety, adherence or follow-up)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Daumit, Principal Investigator — Johns Hopkins University
Locations (1):
- Joseph Gennusa, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will follow National Institute of Mental Health (NIMH) guidelines.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Jerome GJ, Goldsholl S, Dalcin AT, Gennusa Rd JV, Yuan CT, Brown K, Fink T, Minahan E, Wang NY, Daumit GL, Gudzune K. Comparing Implementation Strategies for an Evidence-Based Weight Management Program Delivered in Community Mental Health Programs: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 May 10;12:e45802. doi: 10.2196/45802. PMID 37163331

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: sites
Period: Overall Study
Arm/Group | Enhanced Implementation Intervention | Standard Implementation Intervention
Started | 54; 5 sites | 38; 4 sites
Staff Coach - Started | 11; 5 sites | 9; 4 sites
Staff Coach - Finished | 10; 5 sites | 4; 3 sites
Client With SMI - Started | 43; 5 sites | 29; 4 sites
Client With SMI - Finished | 41; 5 sites | 16; 3 sites
Completed | 51; 5 sites | 20; 3 sites
Not Completed | 3; 0 sites | 18; 1 sites
Not completed — Staff Coach - Left Oranization | 1 | 1
Not completed — Staff Coach - Withdrawal by Site | 0 | 2
Not completed — Staff Coach - Withdrawal by subject | 0 | 1
Not completed — Staff Coach - Lost to follow-up | 0 | 1
Not completed — Client with SMI - Lost to follow-up | 2 | 1
Not completed — Client with SMI - Left organization | 0 | 1
Not completed — Client with SMI - Withdrawal by site | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Implementation Intervention: Client With SMI; Enhanced Implementation Intervention: Staff Coach: The enhanced version will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice as well as organizational strategy meetings. The enhanced version will also include performance coaching.
  training including in-person and online: training, motivational interviewing practice
  organizational strategy meetings: meetings with leadership to optimize implementation of evidence-based practices
  performance coaching: to enhance ability to deliver the weight management intervention
- Standard Implementation Intervention: Client With SMI; Standard Implementation Intervention: Staff Coach: The standard version will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice as well as organizational strategy meetings.
  training including in-person and online: training, motivational interviewing practice
  organizational strategy meetings: meetings with leadership to optimize implementation of evidence-based practices
- Total: Total of all reporting groups
Arm/Group | Enhanced Implementation Intervention: Client With SMI | Enhanced Implementation Intervention: Staff Coach | Standard Implementation Intervention: Client With SMI | Standard Implementation Intervention: Staff Coach | Total
Number analyzed (Participants) | 43 | 11 | 29 | 9 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 11 | 29 | 9 | 89
  >=65 years | 3 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 10 | 18 | 8 | 60
  Male | 19 | 1 | 11 | 1 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 0 | 4
  Not Hispanic or Latino | 42 | 8 | 29 | 9 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 21 | 0 | 13 | 3 | 37
  White | 20 | 10 | 16 | 5 | 51
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 11 | 29 | 9 | 92

OUTCOME MEASURES:

1. Primary Outcome: Knowledge of ACHIEVE Intervention Topics
Description: Knowledge to deliver the intervention using a measure developed by the study team with questions related to weight management and group exercise, 22 questions, each either correct or incorrect. Score range 0-22 will reflect number of questions answered correctly. Higher score indicates better performance.
Time Frame: Baseline and 6 months
Population: Participants from a site that withdrew without implementing the program were not included in analysis models, data was not collected. All participants at sites that delivered the program were analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Enhanced Implementation Intervention- Staff Coach: The enhanced version will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice as well as organizational strategy meetings. The enhanced version will also include performance coaching.
  training including in-person and online: training, motivational interviewing practice
  organizational strategy meetings: meetings with leadership to optimize implementation of evidence-based practices
  performance coaching: to enhance ability to deliver the weight management intervention
- Standard Implementation Intervention- Staff Coach: The standard version will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice as well as organizational strategy meetings.
  training including in-person and online: training, motivational interviewing practice
  organizational strategy meetings: meetings with leadership to optimize implementation of evidence-based practices
Arm/Group | Enhanced Implementation Intervention- Staff Coach | Standard Implementation Intervention- Staff Coach
Number analyzed (Participants) | 11 | 7
score on a scale
  baseline | 16.1 (2.8) | 13.3 (3.5)
  6 months | 19.9 (1.7) | 20.5 (1.4)
Statistical Analysis 1: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; comparison of baseline and 6 months across both groups; Test type: Superiority; Mean Difference (Net) = 5.5, 95% CI 2-sided [3.9 to 7.1]
Statistical Analysis 2: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; between groups differences of change between baseline and 6 months; Test type: Superiority; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.3 to 1.1]

2. Primary Outcome: Self-efficacy to Deliver ACHIEVE Intervention
Description: Self-efficacy to deliver the intervention using a measure developed by the study team with a score range of 1-10. A higher score is better and indicates higher confidence to deliver the intervention.
Time Frame: Baseline and 6 months
Population: Participants from a site that withdrew without implementing the program were not included in analysis models, data not collected. All participants at sites that delivered the program were analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Implementation Intervention- Staff Coach | Standard Implementation Intervention- Staff Coach
Number analyzed (Participants) | 11 | 7
score on a scale
  leading behavioral weight loss group- baseline | 8.9 (0.7) | 9.3 (1.1)
  leading behavioral weight loss group- 6 month | 8.4 (1.4) | 8.9 (0.7)
  completing weigh ins- baseline | 9.0 (1.0) | 9.5 (1.0)
  completing weigh ins- 6 months | 8.1 (1.6) | 9.1 (0.6)
  managing group session- baseline | 9.3 (0.9) | 9.3 (1.1)
  managing group session- 6 months | 8.6 (1.4) | 8.9 (0.9)
Statistical Analysis 1: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; leading behavioral weight loss group baseline to 6 months comparison; Test type: Superiority; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.4 to 0.4]
Statistical Analysis 2: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; leading behavioral weight loss group between group comparison of change; Test type: Superiority; Mean Difference (Net) = -.05, 95% CI 2-sided [-2.0 to 1.0]
Statistical Analysis 3: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; completing weight ins baseline to 6 month comparison; Test type: Superiority; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.4 to 0.2]
Statistical Analysis 4: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; completing weigh ins between groups comparison of change; Test type: Superiority; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.5 to 0.5]
Statistical Analysis 5: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; managing a group session baseline to 6 months comparison; Test type: Superiority; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.2 to 0.3]
Statistical Analysis 6: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; managing a group session between groups comparison of change; Test type: Superiority; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.0 to 1.1]

3. Primary Outcome: Fidelity to ACHIEVE Intervention
Description: Fidelity to the intervention using a tool rating minimal competencies in delivering the intervention. This is a closed ended rating form where coaches are observed and rated. Total scores ranged from 0 to 34 with higher scores indicating higher fidelity.
Time Frame: Baseline (after initial training) and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Implementation Intervention- Staff Coach | Standard Implementation Intervention- Staff Coach
Number analyzed (Participants) | 11 | 7
score on a scale
  baseline | 29.5 (2.9) | 25.5 (3.8)
  6 months | 29.9 (5.9) | 30.7 (2.6)
Statistical Analysis 1: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; comparison between baseline and 6 months across groups; Test type: Superiority; Mean Difference (Net) = 0.5, 95% CI 2-sided [-2.0 to 2.9]
Statistical Analysis 2: Comparison: Enhanced Implementation Intervention- Staff Coach vs Standard Implementation Intervention- Staff Coach; between groups comparison of change post training to 6 months; Test type: Superiority; Mean Difference (Net) = -4.1, 95% CI 2-sided [-9.1 to 0.8]

4. Secondary Outcome: Added Sugar Consumption as Measured by National Health Interview Survey (NHIS) Five Factor Dietary Screener Survey
Description: Participants self reported responses to the NHIS five factor dietary screener. The potential values range from 0 servings to no upper limit with higher numbers indicating higher amounts of food product consumed.
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tsp/day
Groups:
- Enhanced Implementation Intervention- Client With SMI: The enhanced version will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice as well as organizational strategy meetings. The enhanced version will also include performance coaching.
  training including in-person and online: training, motivational interviewing practice
  organizational strategy meetings: meetings with leadership to optimize implementation of evidence-based practices
  performance coaching: to enhance ability to deliver the weight management intervention
- Standard Implementation Intervention- Client With SMI: The standard version will train community mental health program staff to become ACHIEVE-D coaches and peers to become ACHIEVE-D peer-leaders, will include in-person and online training and avatar-assisted motivational interviewing practice as well as organizational strategy meetings.
  training including in-person and online: training, motivational interviewing practice
  organizational strategy meetings: meetings with leadership to optimize implementation of evidence-based practices
Arm/Group | Enhanced Implementation Intervention- Client With SMI | Standard Implementation Intervention- Client With SMI
Number analyzed (Participants) | 43 | 18
tsp/day
  added sugar (tsp/day)- baseline | 20.7 (15.5) | 20.9 (21.0)
  added sugar (tsp/day)- 6 month | 15.0 (10.2) | 20.0 (21.0)
Statistical Analysis 1: Comparison: Enhanced Implementation Intervention- Client With SMI vs Standard Implementation Intervention- Client With SMI; comparison of baseline to 6 months across both groups; Test type: Superiority; Mean Difference (Net) = -3.3, 95% CI 2-sided [-6.9 to 0.3]
Statistical Analysis 2: Comparison: Enhanced Implementation Intervention- Client With SMI vs Standard Implementation Intervention- Client With SMI; comparison of between group differences baseline to 6 months; Test type: Superiority; Mean Difference (Net) = -4.8, 95% CI 2-sided [-11.4 to 1.8]

5. Secondary Outcome: Fruit and Vegetable Consumption as Measured by National Health Interview Survey (NHIS) Five Factor Dietary Screener Survey
Description: as for outcome 4
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: servings/day
Arm/Group | Enhanced Implementation Intervention- Client With SMI | Standard Implementation Intervention- Client With SMI
Number analyzed (Participants) | 43 | 18
servings/day
  Baseline | 3.4 (1.7) | 4.5 (4.1)
  fruit and vegetables (servings/day)-6 months | 3.8 (2.1) | 4.7 (3.0)
Statistical Analysis 1: Comparison: Enhanced Implementation Intervention- Client With SMI vs Standard Implementation Intervention- Client With SMI; Comparison of Baseline & 6 Months across both groups; Test type: Superiority; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.4 to 1.1]
Statistical Analysis 2: Comparison: Enhanced Implementation Intervention- Client With SMI vs Standard Implementation Intervention- Client With SMI; Between Groups Differences of Change between Baseline & 6 Months; Test type: Superiority; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.0 to 0.2]

6. Secondary Outcome: Consumer Sedentary Behavior
Description: CARDIA-EARLY Sedentary Behavior questionnaire. 12-item sedentary behavior measure which separately estimates the amount of time (None,15 minutes or less, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours or more) spent on six categories of sedentary behaviors for an average weekday or weekend day. These responses are then summed to create separate estimates of average weekday and weekend day total sedentary behavior. A weekly estimate of sedentary behavior these scores are weighted and then summed for a total score which ranges from 0 to 168 hours and an average day estimate is calculated by dividing this weekly estimate by 7 (0 to 24).
  Scores reported below reflect the average day estimate of sedentary behavior with a possible score range of 0 to 24 hours. For all scoring a higher score indicates more sedentary activity completed in the day. Higher score is worse.
Time Frame: Baseline and 6 months
Population: Participants from a site that withdrew without implementing the program were not included in analysis models, data not colleccted. All participants at sites that delivered the program were analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Enhanced Implementation Intervention- Client With SMI | Standard Implementation Intervention- Client With SMI
Number analyzed (Participants) | 43 | 18
hours/day
  Baseline | 8.9 (5.9) | 11.0 (7.4)
  6 Month | 7.9 (6.6) | 8.5 (5.3)
Statistical Analysis 1: Comparison: Enhanced Implementation Intervention- Client With SMI vs Standard Implementation Intervention- Client With SMI; comparison of between group differences baseline to 6 months; Test type: Superiority; Mean Difference (Net) = -0.6, 95% CI 2-sided [-4.5 to 3.3]
Statistical Analysis 2: Comparison: Enhanced Implementation Intervention- Client With SMI vs Standard Implementation Intervention- Client With SMI; comparison of baseline to 6 months across groups; Test type: Superiority; Mean Difference (Net) = -1.6, 95% CI 2-sided [-3.1 to 0.2]

7. Secondary Outcome: Client Weight
Description: Weight measured in kilograms (kg) using a calibrated scale and standardized procedures
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Enhanced Implementation Intervention- Client With SMI | Standard Implementation Intervention- Client With SMI
Number analyzed (Participants) | 43 | 18
kg
  baseline | 111.9 (27.2) | 114.8 (28.2)
  6 months | 106.5 (27.3) | 112.7 (30.5)
Statistical Analysis 1: Comparison: Enhanced Implementation Intervention- Client With SMI vs Standard Implementation Intervention- Client With SMI; comparison of baseline and 6 months across groups; Test type: Superiority; Mean Difference (Net) = -3.8, 95% CI 2-sided [-6.1 to -1.6]
Statistical Analysis 2: Comparison: Enhanced Implementation Intervention- Client With SMI vs Standard Implementation Intervention- Client With SMI; between groups differences of change between baseline to 6 months; Test type: Superiority; Mean Difference (Net) = -6.6, 95% CI 2-sided [-20.2 to 6.9]

8. Secondary Outcome: Continued Site Implementation
Description: Sites reported whether program was still being delivered six months after original study period.
Time Frame: 12 months (6 months after original study period of Baseline to 6 months)
Population: A site that withdrew without implementing the program could not be included in the analysis of continued site implementation.
Measure: Number; unit: sites
Units Other Than Participants: Sites
Arm/Group | Enhanced Implementation Intervention | Standard Implementation Intervention
Number analyzed (Participants) | 11 | 7
Number analyzed (Sites) | 5 | 3
sites
  Implementing after 6 months | 4 | 0
  Not implementing after 6 months | 1 | 3

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Description: Adverse events were only collected for Client participants with serious mental illness who were participating in the study.
Arm/Group | Enhanced Implementation Intervention | Standard Implementation Intervention
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/29
Serious Adverse Events (participants affected / at risk) | 3/43 | 3/29
Other Adverse Events (participants affected / at risk) | 4/43 | 1/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Implementation Intervention (N=43) | Standard Implementation Intervention (N=29)
mental health hospitalization (Psychiatric disorders) | 2 (2) | 1 (1)
infection treatment (Infections and infestations) | 1 (1) | 2 (2)
spinal injection (Surgical and medical procedures) | 1 (1) | 0 (0)
head injury (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Implementation Intervention (N=43) | Standard Implementation Intervention (N=29)
outpatient procedure (Surgical and medical procedures) | 3 (3) | 1 (1)
accident or injury (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03454997/Prot_SAP_000.pdf